CLINICAL TRIAL: NCT07194941
Title: Efficacy and Safety of Fecal Microbiota Transfer (FMT) for Recurrent Urinary Tract Infections in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEMINALE-II
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Urinary Tract Infections in Women
Keywords: Women; Urinary tract infections; Fecal microbiota
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total dose of 150 g of fresh feces (Experimental): 150 g freeze-dried product of fresh feces (~30 capsules) to be taken throughout the day.
  Interventions: Biological: Freeze-dried product made of fresh feces
- Total dose of 300 g of fresh feces (Experimental): Freeze-dried product made from 150 g of fresh feces (~30 capsules) to be taken throughout the day. Subsequently, for 15 days (2 capsules per day in a single dose) made from 150 g of fresh feces. Receiving a total dose of 300 g of fresh feces.
  Interventions: Biological: Freeze-dried product made of fresh feces

INTERVENTIONS:
Biological: Freeze-dried product made of fresh feces — FMT represents an ecological alternative for restoring the damaged intestinal ecosystem in this infection, increasing ecological diversity and thus limiting the spread of the pathogen. Recurrence of C. difficile is its only approved indication.
  The impact of FMT on the intestinal ecosystem is attributable to intraspecific bacterial competition: commensal microorganisms (sensitive and non-virulent) have more effective growth rates than pathogenic bacteria (resistant and virulent), so FMT produces an ecological replacement in favor of grafting the donor microbiota and eliminating antibiotic-resistant clones.

SUMMARY:
Urinary tract infections (UTIs) are highly prevalent worldwide, especially in women, with frequent recurrences and significant healthcare costs. The proposed Phase II clinical trial will define dosing and administration strategies for FMT in recurrent UTIs. If effective, this ecological approach could provide a novel therapeutic alternative to antibiotics for one of the most common infectious diseases worldwide

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are highly prevalent worldwide, especially in women, with frequent recurrences and significant healthcare costs. Current treatment relies mainly on antibiotics, which contribute to antimicrobial resistance and adverse effects. While preventive strategies such as antibiotic prophylaxis, personalized vaccines, D-mannose, or hyaluronic acid instillations have been explored, they show limited success, partly because the intestinal tract acts as the reservoir for uropathogens.

This project proposes fecal microbiota transplantation (FMT) from healthy donors to modify the intestinal microbiome of patients with recurrent UTIs, aiming to eradicate intestinal colonization by resistant pathogens and prevent urinary infections. FMT, already approved for recurrent Clostridioides difficile since 2015, has evolved from colonoscopy-based procedures to oral capsules. Observations in clinical practice suggest FMT may incidentally clear recurrent UTIs and multidrug-resistant bacteria, though no formal indication exists yet due to lack of evidence on optimal dose and regimen.

The proposed Phase II clinical trial will define dosing and administration strategies for FMT in recurrent UTIs. If effective, this ecological approach could provide a novel therapeutic alternative to antibiotics for one of the most common infectious diseases worldwide

ELIGIBILITY:
Inclusion Criteria:

Women ≥18 years of age with UTIs (≥3 episodes in one year or ≥2 in six months) who meet at least one of the following criteria

* UTIs despite having used other prophylactic strategies.
* HUTI due to resistant bacteria (ESBL- or carbapenemase-producing Enterobacteriaceae, and quinolone-resistant Pseudomonas aeruginosa or Enterococcus faecium).
* Allergy or previous adverse reactions to available oral antibiotics (usually beta-lactams, but could occur with other antibiotic families) for prophylaxis and/or treatment.

Exclusion Criteria:

* Have symptoms compatible with symptomatic UTI at the time of inclusion or be undergoing treatment for it.
* Be receiving another preventive strategy for UTIs at the time of study inclusion: prophylactic antibiotics, bladder instillation with hyaluronic acid, D-mannose, or therapeutic vaccines. In the case of the latter, Version 3.0_ March 22, 2023 13 patients who have received them must have had at least two recurrences despite their administration.
* Rifaximin allergy.
* Inability to understand the study and sign the informed consent form, and to collect stool and urine samples.
* Pregnancy or breastfeeding
* Patients with bone marrow or solid organ transplants (patients who have been transplanted for ≥ 5 years and are stable from a transplant perspective are allowed to be included).
* Any clinically significant disease at the investigator's discretion, other than UTIs, that is not medically controlled at the time of study inclusion.
* Patients with lithiasis or permanent catheters (patients with self-catheters are excluded).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Assess the usefulness of TMF in preventing episodes of ITUr. | 12 months
  Proportion (%) of patients free of ITUr 12 months after the start of the study.

SECONDARY OUTCOMES:
To evaluate the efficacy of two different TMF dosages in modifying the microbiota and achieving a reduction in the frequency of episodes in patients with rUTI. | 12 months
  Proportion of patients recurrence-free at 12 months (%)
To evaluate the efficacy of two different TMF dosages in modifying the microbiota and achieving a reduction in the frequency of episodes in patients with rUTI. | 12 months
  Recurrence-free time (days)
To evaluate the efficacy of two different TMF dosages in modifying the microbiota and achieving a reduction in the frequency of episodes in patients with rUTI. | 12 months
  Time between recurrences (days)
To evaluate the efficacy of two different TMF dosages in modifying the microbiota and achieving a reduction in the frequency of episodes in patients with rUTI. | 12 months
  Annual recurrence rate (number of recurrences per patient per year, additional clinical information such as whether the symptoms are more like cystitis or pyelonephritis, and the need for hospital admission).
Tolerability and safety of FMT | 12 months
  Proportion of the following adverse reactions: diarrhoea, abdominal pain, nausea, fever, low-grade fever, abdominal distension, vomiting, constipation, flatulence, rectal bleeding, skin rash, others).
FMT impact on intestinal bacterial ecosystem | 12 months
  Document clonal replacement in classical cultivable bacteria and demonstrate the impact of FMT on the entire intestinal bacterial ecosystem through next-generation sequencing of the 16S rDNA gene and metabolic monitoring by determining short-chain fatty acids.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Soriano, MD, Principal Investigator — HOSPITAL CLINIC DE BARCELONA, SPAIN; Antonio Ramos, MD, Principal Investigator — HOSPITAL UNIVERSITARIO PUERTA DE HIERRO, MADRID, SPAIN; Luis Llanes, MD, Principal Investigator — HOSPITAL UNIVERSITARIO DE GETAFE, MADRID, SPAIN
Locations (1):
- IRyCIS - FIBIO Hospital Ramón y Cajal, Madrid, Spain